CLINICAL TRIAL: NCT03046680
Title: Health Coaching Based Treatment Versus Usual Treatment of Systemic Arterial Hypertension and Comorbidities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Principal Investigator, Sayuri Inuzuka, Cardiologist, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFGoias
Record Dates: First submitted 2017-02-01; First posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Hypertension, Resistant to Conventional Therapy
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Coaching (Experimental): Individualized follow-up, supporting the individual for a better autonomy in personal care.
  Interventions: Other: Health Coaching
- Multiprofessional Team (Active Comparator): Physician, nurse, nutrionist usual care.
  Interventions: Other: Multiprofessional Team

INTERVENTIONS:
Other: Health Coaching
  Arms: Health Coaching
Other: Multiprofessional Team
  Arms: Multiprofessional Team

SUMMARY:
Hypertension is a multifactorial clinical condition, it may not cause symptoms and its diagnosis is often delayed. And even when it is diagnosed early, some patients cannot manage an adequate blood pressure.

There are several hypotheses for the non-control of blood pressure, among them the difficulty of lifestyle change, irregular treatment with antihypertensive drugs, non-individualized treatment. Studies haven shown that tools such as multiprofessional team and hypertension leagues are important strategies to obtain a better outcome in the hypertension treatment, but new approaches are still necessary. Health Coaching is an individualized form of follow-up, promoting better adherence, better nutrition, smoking cessation, regular physical exercise and regular use of drugs, thus reducing cardiovascular mortality.

DETAILED DESCRIPTION:
Drug adherence and lifestyle changes are tools for chronic disease control. The relationship between nutrients, alcohol intake, and weight change in blood pressure was demonstraded in one study, demonstrating the importance of lifestyle change. Studies have shown that multiprofessional team and hypertension leagues are important strategies to obtain a better outcome, but new approaches to the patient are still necessary. Health coaching is an individualized follow-up, promoting better adherence to the hypertension treatment. Health coaching is a new model based on the support of the individual, for a better autonomy in personal care. The process engages de patient with the conditions of the disease itself by increasing knowledge, skill and confidence so that the patient become informed, active in the participation of its own care. Among health care, training is characterized by the expression. Of concerns, answering questions, providing information on home-based follow-up, and collaborative development of health care plans.

Motivated patients are more likely to treatment adherence and more committed to making lifestyle changes and thus effectively managing their illness.

The research is a randomized clinical trial comparing treatment based on health coaching and the usual treatment based in the treatment of hypertension and comorbidities in uncontrolled hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Blood pressure above 160/90mmHg
* Signed the free and informed consent form
* Regularly enrolled, with at least two visits in the last 12 months

Exclusion Criteria:

* Miss the subsequent consultation
* Those who have not signed the free informed consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-06-01 (Estimated); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Grade 2 hypertension achieving blood pressure control (Graded According to NCI CTCAE Version 3.0) | 6 months
  Number of patients with grade 2 hypertension reaching BP <140 / 90mmHg.
Lifestyle Changes | 6 months
  Number of patients with grade 2 hypertension who were able to lose weight, adhere to physical exercises, reduce dietary salt.
Treatment Adhesion | 6 months
  Number of patients with grade 2 hypertension who took the drugs according to the medical prescription

CONTACTS AND LOCATIONS:
Overall Officials: Thiago Veiga Jardim, Study Chair — Universidade Federal de Goias
Locations (1):
- Universidade Federal de Goias, Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: Undecided